CLINICAL TRIAL: NCT06888609
Title: Comparison of Back Extensor Strengthening Versus Core Stability Exercise in Patients With Thoracic Kyphosis
Brief Title: Comparing Back Extensor and Core Stability Training in Kyphosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-01003 Zahoor Ahmad
Record Dates: First submitted 2025-02-20; First posted 2025-03-21 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-04

CONDITIONS: Thoracic Kyphosis
Keywords: Posture; Spinal Alignment; Overall Functional Outcome; Pain; Range of Motion
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation; Analgesia; Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Back Extensor Strengthening Exercises (Experimental): Usage of modalities like hot pack & TENS along with certain exercises mentioned in the following:
  1. Superman Exercise (Prone position, lift chest off ground, arms extended)
  2. Prone Arm and Leg Raise (Prone, lift opposite arm & leg)
  3. Seated Row (Resistance Band) (Pull band towards chest)
  4. Wall Angels (Standing against wall, moving arms up/down)
  Interventions: Other: Back Extensor Strengthening Exercises
- Core Stability Exercises (Experimental): Usage of modalities like hot pack & TENS along with certain exercises mentioned in the following:
  1. Side Plank (Side-lying, lift hips while maintaining straight posture)
  2. Dead Bug Exercise (Supine, extend opposite arm & leg)
  3. Bridging Exercise (Supine, lift hips to straight line)
  4. Bird-Dog Exercise (Quadruped, extend opposite arm & leg)
  Interventions: Other: Core Stability Exercises

INTERVENTIONS:
Other: Back Extensor Strengthening Exercises — 1. Superman Exercise Sets/Reps: 2 sets × 10-12 reps, hold 5-10 sec
  2. Prone Arm and Leg Raise Sets/Reps: 2 sets × 10-12 reps, hold 5-10 sec
  3. Seated Row (Resistance Band) Sets/Reps: 2 sets × 12-15 reps, hold 3-5 sec
  4. Wall Angels Sets/Reps: 2 sets × 10-12 reps, 3-5 sec per cycle
  Other Names: Hot Pack (15-20 mins) - Upper back & thoracic spine for relaxation; TENS (10 mins)- Applied to thoracic region for pain relief (Before & after exercises)
  Arms: Back Extensor Strengthening Exercises
Other: Core Stability Exercises — 1. Side Plank Sets/Reps: 3 sets, hold 10-60 sec per side
  2. Dead Bug Exercise Sets/Reps: 3 sets × 6-15 reps per side
  3. Bridging Exercise Sets/Reps: 3 sets × 10-20 reps, hold 2-5 sec
  4. Bird-Dog Exercise Sets/Reps: 3 sets × 8-15 reps per side, hold 2-5 sec
  Other Names: Hot Pack (15-20 mins) - Upper back & thoracic spine for relaxation; TENS (10 mins)- Applied to thoracic region for pain relief (Before & after exercises)
  Arms: Core Stability Exercises

SUMMARY:
To compare the effects of back extensor strengthening exercises versus core stability exercises on thoracic kyphosis in patients, assessing improvements in posture, spinal alignment, and overall functional outcomes

DETAILED DESCRIPTION:
Kyphosis is the normal forward curvature of our spine and when this curvature becomes excessively increased is referred to as hyper kyphosis or Hunch back. Its normal value is between 20 and 40 degrees. When the thoracic kyphotic angle exceeds 40 degrees, it is referred to as hyper kyphosis. The three main types of kyphosis often seen in individuals are postural, Structural and congenital. Postural kyphosis is caused by high external load on individual spine having overall poor muscle strength. Sagittal misalignment can be caused by poor posture while sitting and standing as well as prolonged sitting.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-40 years with a diagnosis of mild to moderate thoracic kyphosis (Cobb angle between 40° and 60°).
* The presence of back pain or discomfort is attributed to kyphosis.
* Willingness to participate and commit to the study's duration (6 weeks of intervention and follow-up).
* Ability to provide informed consent.

Exclusion Criteria:

* Severe thoracic kyphosis (Cobb angle > 60°).
* Other spinal conditions such as scoliosis or spinal fractures.
* Previous spinal surgery or contraindications to physical activity.
* Neurological disorders affecting motor function.
* Pregnancy or severe medical comorbidities that would preclude participation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity Measured by Visual Analogue Scale (VAS) | 12 Weeks
  A 10 cm horizontal line with "No Pain" (0) on the left and "Worst Pain" (10) on the right. Patients mark their pain level on the scale before and after interventions to assess changes. Test-Retest Reliability: The VAS shows high test-retest reliability, especially in literate populations (r = 0.94), indicating stable pain scores over time when used with the same individual. Validity effectively captures the full spectrum of pain intensity, making it a valid tool for assessing the pain experience of thoracic kyphosis patients.
Change in Thoracic Spine Range of Motion (ROM) Measured by Inclinometer | 12 Weeks
  The inclinometer has demonstrated good test-retest reliability, with high correlation (r = 0.90) in measuring range of motion (ROM) over time when used consistently on the same patient.The inclinometer accurately measures thoracic spine mobility and is considered a valid tool for assessing movement restriction or improvement in patients with thoracic kyphosis.
Assessment of Postural Deformity Severity Using the Matthias Test | 12 Weeks
  It is effective in identifying postural deformities and the severity of thoracic kyphosis. The Matthias Test has demonstrated good inter-rater reliability.
Change in Disability Level Measured by Oswestry Disability Index (ODI) | 12 Weeks
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability.
Change in Functional Disability Measured by Roland-Morris Disability Questionnaire (RDQ) | 12 Weeks
  The Roland-Morris Disability Questionnaire is most sensitive for patients with mild to moderate disability due to acute, sub-acute, or chronic low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Sadiq, MSPT (OMPT), Principal Investigator — Riphah International University
Locations (1):
- DHQ Timergara & Batkhela, Malakand, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No